CLINICAL TRIAL: NCT05875168
Title: Phase 1/2, Open-label, Multicenter, First-in-Human Study of DS-3939a in Subjects With Advanced Solid Tumors
Brief Title: First-in-Human Study of DS-3939a in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DS3939-077
Record Dates: First submitted 2023-05-10; First posted 2023-05-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: DS-3939a; anti-body drug conjugate; advanced/metastatic solid tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Part 1) (Experimental): Participants with locally advanced, metastatic, or unresectable tumors who will receive an intravenous (IV) infusion of DS-3939a.
  Interventions: Drug: DS-3939a
- Dose Expansion (Part 2) (Experimental): Multiple expansion cohorts targeting various advanced solid tumors.
  Interventions: Drug: DS-3939a

INTERVENTIONS:
Drug: DS-3939a — One IV infusion Q3W on Day 1 of each 21-day cycle

SUMMARY:
This study will evaluate the safety, tolerability, and efficacy of DS-3939a in participants with advanced solid tumors.

DETAILED DESCRIPTION:
DS-3939a is an antibody drug conjugate (ADC) being developed for the treatment of malignant tumors. This is a first-in-human, dose-escalating clinical study divided into 2 parts: the Dose Escalation Part (Part 1) and the Dose Expansion Part (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Sign and date the main Informed Consent Form (ICF).
* Has a left ventricular ejection fraction ≥50% by either an echocardiogram or multigated acquisition within 28 days of enrollment.
* Has adequate organ function.
* Measurable disease based on RECIST V1.1.
* Eastern Cooperative Oncology Group performance status score of 0 or 1.

Additional inclusion criteria for Part 1

* Has a histologically or cytologically documented locally advanced, metastatic, or unresectable solid malignant tumors.

Additional inclusion criteria for Part 2

* Has a histologically or cytologically documented locally advanced, metastatic, or unresectable cancer meeting the protocol criteria and documented radiographic disease progression during or after the most recent anticancer therapy.
* Is able to provide either of the following baseline tumor samples:

  * Fresh tumor biopsy samples meeting either of the following requirements that were obtained during the Main Screening or Tissue Screening Period, or
  * Fresh core needle biopsy sample
  * Biopsy samples obtained with forceps or cryobiopsy, such as bronchoscopic or transbronchial lung biopsy (if the sample amount is equivalent to core needle biopsy and processing after sample collection follows the procedure described in the Study Laboratory Manual)
  * FFPE tumor tissue samples obtained by biopsy or surgery performed within 6 months before signing the main ICF. If samples were obtained prior to the start of the most recent anticancer therapy, the Sponsor Medical Monitor should be consulted regarding the adequacy of the sample.

Exclusion Criteria:

* Has had prior treatment targeting mucin 1 (MUC1) or TA-MUC1.
* Has spinal cord compression or clinically active central nervous system metastases.
* Has multiple primary malignancies, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated, with no evidence of disease for ≥3 years.
* Has a history of noninfectious interstitial lung disease (ILD)/pneumonitis (including suspected one), has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
* Has active or uncontrolled human immunodeficiency virus (HIV) infection.
* Has evidence of active or uncontrolled hepatitis B virus or hepatitis C virus infection.
* Any of the following within the past 6 months: cerebrovascular accident, transient ischemic attack, or other arterial thromboembolic event.
* Has an active, known, or suspected autoimmune disease.
* Current participation in other therapeutic investigational procedures, except for participation in Long Term Follow-Up without any investigational treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2027-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities Following Treatment With DS-3939a | Approximately 3 months after first dosing
Overall Number of Participants with Treatment-emergent Adverse Events and Serious Adverse Events Following Treatment With DS-3939a | Up to approximately 31 months
Number of Participants with Objective Response Rate Following Treatment With DS-3939a (Part 2) | Up to approximately 31 months

SECONDARY OUTCOMES:
Number of Participants with Objective Response Rate Following Treatment With DS-3939a (Part 1) | Up to approximately 31 months
Disease Control Rate Following Treatment With DS-3939a | Up to approximately 31 months
Duration of Response Following Treatment With DS-3939a | Up to approximately 31 months
Time to Response Following Treatment With DS-3939a | Up to approximately 31 months
Progression Free Survival Following Treatment With DS-3939a | Up to approximately 31 months
Overall Survival Following Treatment With DS-3939a | Up to approximately 31 months
TA-MUC1 Expression by Immunohistochemistry Following Treatment With DS-3939a | At Cycle 1 Day 1
Area Under the Plasma Concentration Curve (AUC) Following Treatment With DS-3939a | Cycles 1 & 3: Days 1, 2, 4, 8 & 15; Cycle 2: Day 1 & 1 time between Days 3 to 8 (Part 2 Only); Cycles 4 & every 2 cycles thereafter up to 31 months: Day 1 (each cycle is 21 days)
Maximum Plasma Concentration (Cmax) Following Treatment With DS-3939a | Cycles 1 & 3: Days 1, 2, 4, 8 & 15; Cycle 2: Day 1 & 1 time between Days 3 to 8 (Part 2 Only); Cycles 4 & every 2 cycles thereafter up to 31 months: Day 1 (each cycle is 21 days)
Time to Maximum Plasma Concentration (Tmax) Following Treatment With DS-3939a | Cycles 1 & 3: Days 1, 2, 4, 8 & 15; Cycle 2: Day 1 & 1 time between Days 3 to 8 (Part 2 Only); Cycles 4 & every 2 cycles thereafter up to 31 months: Day 1 (each cycle is 21 days)
Minimum Observed Concentration (Ctrough) Following Treatment With DS-3939a | Cycles 1 & 3: Days 1, 2, 4, 8 & 15; Cycle 2: Day 1 & 1 time between Days 3 to 8 (Part 2 Only); Cycles 4 & every 2 cycles thereafter up to 31 months: Day 1 (each cycle is 21 days)
Terminal Half-Life (T1/2) Following Treatment With DS-3939a | Cycles 1 & 3: Days 1, 2, 4, 8 & 15; Cycle 2: Day 1 & 1 time between Days 3 to 8 (Part 2 Only); Cycles 4 & every 2 cycles thereafter up to 31 months: Day 1 (each cycle is 21 days)
Number of Participants With Treatment-emergent Anti-drug Antibodies Following Treatment With DS-3939a | Up to approximately 47 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (32):
- United States (6):
  - Florida Cancer Specialists, Sarasota, Florida
  - Oregon Health & Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - The Medical College of Wisconsin, INC, Milwaukee, Wisconsin
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - McGill University Health Center, Montreal
  - Princess Margaret Cancer Center, Toronto
- China (4):
  - Beijing Cancer Hospital, Beijing
  - Shandong Cancer Hospital, Jinan
  - The Second Peoples Hospital of Neijiang, Neijiang
  - Shanghai East Hospital, Shanghai
- France (5):
  - Centre Léon Bérard, Lyon
  - Assistance Publique- de Marseille, Marseille
  - Chu Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Japan (5):
  - National Cancer Center Hospital, Chūōku
  - Kansai Medical University Hospital, Hirakata-shi
  - National Cancer Center Hospital East, Kashiwa
  - Cancer Institute Hospital of Jfcr, Kōtoku
  - Kindai University Hospital, Ōsaka-sayama
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Next Madrid, Pozuelo de Alarcón
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Takano K, Yukiura M, Takahashi K, Kitamura M, Okuno H, Shiose Y, Honda K, Oyama K, Yamada M, Obuchi W, Kumagai K, Sakurai K, Goto R, Zembutsu A, Kagari T, Abe Y, Agatsuma T. DS-3939a: A TA-MUC1-Directed Antibody-Drug Conjugate with Broad Antitumor Activity. Mol Cancer Ther. 2026 Jan 2;25(1):7-20. doi: 10.1158/1535-7163.MCT-24-0666. PMID 40635151